CLINICAL TRIAL: NCT01831323
Title: Evaluation of the Metabolome in Diverticular Disease and Effects of Probiotic Mixture VSL#3 vs Fibers, Rifaximin and Mesalazine on the Metabolome in Diverticular Disease of the Colon
Brief Title: Evaluation of the Metabolome in Diverticular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: S.Eugenio Hospital (Other)
Responsible Party: Principal Investigator, Gian Marco Giorgetti, Dott. in Medicina Interna, Chirurgia oncologica, immunologia e allergologia, S.Eugenio Hospital
Other Study IDs: TUR-SUDD 2012
Record Dates: First submitted 2012-12-04; First posted 2013-04-15 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Simple Diverticular Disease
MeSH Terms: interventions — Rifaximin; Mesalamine; Anti-Inflammatory Agents; Psyllium

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine and stools
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- mesalazine: 10 female patients with first diagnosis of SUDD will take mesalazine 1,6g per day for 14 days (1 tablet 800mg twice daily)
  Interventions: Drug: Mesalazine
- VSL#3: 10 female patients with first diagnosis of SUDD will take VSL#3 2 sachets a day for 14 days (1 sachet twice a day, for a total of 900 billion bacteria per day)
  Interventions: Dietary Supplement: VSL#3
- Rifaximin: 10 female patients with first diagnosis of SUDD will take 800mg/day of rifaximin (2 tablets of 200mg twice a day)
  Interventions: Drug: Rifaximin
- fiber: 10 female patients with first diagnosis of SUDD will take fibers for 14 days (psyllium 10grams per day)
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: VSL#3 — VSL#3
  Other Names: Probiotic food supplement
  Groups: VSL#3
Drug: Rifaximin — Rifaximin
  Other Names: Unabsorbable antibiotic
  Groups: Rifaximin
Drug: Mesalazine — Mesalazine
  Other Names: anti-inflammatory drug
  Groups: mesalazine
Dietary Supplement: Psyllium — psyllium
  Other Names: Fibers
  Groups: fiber

SUMMARY:
To evaluate the effect of the probiotic formulation VSL#3 on the metabolome and microbiota of diverticular disease, comparing it with the effects exerted by supplementation with fibers, by rifaximin and by mesalazine, and assessing the evolution over time after each specific treatment

DETAILED DESCRIPTION:
The incidence of diverticular disease of the colon has increased over the last few years. Since it presents potentially severe complications (both in terms of morbidity and mortality), the most recent studies are focusing on the underlying mechanisms and therapeutic options.

Diverticular disease of the colon presents important etiopathogenetic events. The first is that the severity of microscopic inflammation is correlated to the disease activity. The second is the bacterial overgrowth which is observed in the colon, where the diverticula form "recesses" where bacteria can proliferate. The third is that the "metabolome" plays an important role in the pathogenesis of diseases of the gastrointestinal tract (and not only). An extensive combination of microbial species live permanently in the human gut and participate in the metabolic activities of the gastro-intestinal tract (such as the synthesis of certain vitamins, improvement of the immune system, and balance of the resident bacterial species). There is little published clinical evidence suggesting a direct link between microbiota and diverticular disease; however, an altered microbiota in the flora of patients with colon cancer, irritable bowel syndrome, and IBD has been described.

It is clear that human metabolism and inflammatory response are influenced by genetic information outside our genome. Insights into the influence of microorganisms on the pathogenesis in gastrointestinal function and diverticular disease are in their infancy and often rely on extrapolation from other disease states. Microbiological analysis of fecal microbiota can provide important information on the role that the microbial-mammalian axis might have on the pathogenesis of diverticular disease.

Alteration of the metabolome play an important role in some pathologies of the gastrointestinal tract, from Inflammatory Bowel Diseases (IBD) to Irritable Bowel Syndrome (IBS). Most likely, it plays the same role in diverticular disease. In fact, the current western diet is poor in fibers and can cause an alteration of the resident bacterial species, with a reduction of bifidobacteria and an increase of clostridia.

This alteration might be present in diverticular disease and the manipulation of the microbial flora might represent both a treatment option for diverticular disease and the prevention of its complications.

Recent studies showed that the treatment with probiotics can help reduce the activity index in patients with DDS and as well as reduce the recurrence of the disease.

A new method has now been validated to assess the microbiota: the analysis of the faecal and urinary metabolome by high resolution Nuclear Magnetic Resonance (NMR) spectroscopy. The microbioma is the combination of the DNA of the microorganisms that compose the intestinal microflora (microbiota). Metabolomics allow to assess the metabolic activity of the microbiota and its possible interactions with the host.

The metabolomic analyses of stools and urine offer a new approach to evaluate the metabolome of diverticular disease, and compare it in patients who take a probiotic, fibers, non-absorbable antibiotics or an anti-inflammatory drug.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age
* Patient with a diagnosis of uncomplicated symptomatic diverticular disease diagnosed for the first time
* Patient able to comply with the procedures of the Protocol
* Ability to sign written informed consent

Exclusion Criteria:

* Segmental colitis associated with diverticulosis
* Inflammatory Bowel Disease
* Active or recent peptic ulceration
* Chronic renal failure
* Known allergy to products in the study
* Use of lactulose-lactitol in the two weeks prior to enrollment and during the study
* Previous surgery of the colon
* Diverticular disease-related complications (fistulas, abscesses, stenosis)
* Use of probiotics in the 4 weeks prior to enrolment
* Renal, hepatic, hematologic, cardiovascular, pulmonary, neurological, psychiatric, immunological, gastrointestinal or endocrine disease, if found to be clinically significant
* Active malignancy or history of any type of malignancy.
* Recent history or suspicion of abuse of alcohol or drugs
* Women who are pregnant, nursing or of childbearing age not using appropriate contraceptive methods
* Any severe pathology that may interfere with the treatment
* Inability to provide written informed consent
* Not sufficiently reliable or presence of conditions that can result in non-compliance / patient adherence to the Protocol
* Previous participation in another study
* Lack of compliance towards the products in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with first diagnosis of uncomplicated symptomatic diverticular disease
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
identify the metabolome of symptomatic uncomplicated Diverticular Disease (SUDD) | 12 months
  As no studies have ever been conducted or published on this aspect, the main outcome of the study is to analyze and identify the metabolome of patients with SUDD before starting any therapy and after a 2 week therapy of a probiotic, fibers or antibiotics. The metabolomic analysis will allow a precise evaluation of the systemic and organ-specific processes based on low molecular weight components thus providing a profile of the metabolic system of these patients.
verify changes in the intestinal microbiota following treatment in the different study groups. | 12 months

SECONDARY OUTCOMES:
evaluate the symptomatology and metabolome | 12 months
  Evaluate the difference in symptomatology in the different groups, in particular stool frequency, abdominal pain, mucus or blood in faeces, intestinal gas, and assess possible link to the different metabolome and microbiota
evaluate the different metabolomes and microbiota according to the treatment used | 12 months
  Evaluate if the variation in metabolome and microbiota induced by the different treatments modify the symptomatology of the patients and for how long.
Evaluate the effects of supplementation with VSL#3 on the metabolome and microbiota of Diverticular Disease | 12 months
  Evaluate the effects of supplementation with VSL#3 on the metabolome and microbiota of Diverticular Disease, comparing it with the effects of supplementation with fibers, or treatment with rifaximin or with mesalazine.
evaluate if difference in the symptomatology in the different groups are correlated with changes in the intestinal microbiota | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gianmarco Giorgetti, Principal Investigator — Sant'Eugenio Hospital
Locations (1):
- Sant'Eugenio Hospital, Rome, RM, Italy